CLINICAL TRIAL: NCT06969664
Title: A Phase I Clinical Study to Evaluate Effect of High-Fat Diet on Pharmacokinetics of a Single Oral Dose of SHR7280 Tablets and to Assess the Effect of SHR7280 on QT Interval in Healthy Subjects
Brief Title: A Trial of SHR7280 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SHR7280-107
Record Dates: First submitted 2025-05-06; First posted 2025-05-14 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Endometriosis; Uterine Fibroids; Assisted Reproduction
MeSH Terms: conditions — Endometriosis; Leiomyoma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group A (Experimental)
  Interventions: Drug: SHR7280 Tablet; Drug: SHR7280 Placebo Tablet
- Treatment group B (Experimental)
  Interventions: Drug: SHR7280 Tablet; Drug: SHR7280 Placebo Tablet

INTERVENTIONS:
Drug: SHR7280 Tablet — Oral SHR7280 tablet.
Drug: SHR7280 Placebo Tablet — Oral SHR7280 placebo tablet.

SUMMARY:
The study is being conducted to evaluate the effect of high-fat meal on pharmacokinetics of SHR7280 after oral administration and the effect of SHR7280 on QT interval at low and high doses in healthy Chinese volunteers.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily sign the informed consent form prior to any activities in the trail, demonstrate comprehension of the trial procedures and methodology, and agree to strictly adhere to the protocol throughout the study period.
2. Be aged between 18 and 45 years inclusive (determined at the time of signing the informed consent form).
3. Have a body weight of ≥50 kg for males and ≥45 kg for females, with a Body Mass Index (BMI) between 18 and 26 kg/m² inclusive.
4. Have no plans for pregnancy or sperm/egg donation from the time of signing the inform consent form until 1 week after the last administration of the investigational product, and agree to use highly effective contraceptive measures.

Exclusion Criteria:

1. Individuals with a history of chronic or serious diseases, or current conditions affecting the respiratory, circulatory, digestive, urinary, hematological, endocrine, immune, nervous, or psychiatric systems, and deemed ineligible to participate in this trial by the investigator.
2. Females who are pregnant, breastfeeding, or with a positive serum pregnancy test during the screening or baseline period.
3. History of smoking (average daily cigarette consumption >5 cigarettes) within 3 months prior to randomization, or any use of tobacco products during the study period.
4. History of drug abuse, positive urine drug abuse screen at the screening period.
5. Receipt of live (attenuated) vaccines within 1 month prior to screening or planned administration during the trial (excluding influenza vaccines).
6. Undergoing any surgical procedure within 3 months prior to randomization, incomplete recovery from surgery, or anticipated need for surgery or hospitalization during the trial period.
7. Inability to comply with standardized dietary requirements, intolerance to high-fat meals, or presence of dysphagia.
8. Any condition judged by the investigator to potentially affect drug absorption, distribution, metabolism, or excretion, reduce compliance, or pose other risks that make participation in the study inappropriate.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2025-05-19 (Actual); Primary Completion 2025-07-05 (Actual); Study Completion 2025-07-05 (Actual)

PRIMARY OUTCOMES:
Peak concentration (Cmax) | Day 1 to Day 8.
Area under the plasma concentration-time curve from time 0 to the last quantifiable timepoint (AUC0-t) | Day 1 to Day 8.
Area under the plasma concentration-time curve from time 0 to infinity (AUC0-∞) | Day 1 to Day 8.

SECONDARY OUTCOMES:
Time to peak concentration (Tmax) | Day 1 to Day 8.
Elimination half-life (t1/2) | Day 1 to Day 8.
Adverse events (AEs) | Day 1 to Day 15.

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen Memorial Hospital, Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided